CLINICAL TRIAL: NCT05088460
Title: A Randomized Double-Blind Placebo-Controlled Study of the LEPR Agonist Antibody REGN4461 for the Treatment of Metabolic Abnormalities in Patients With Familial Partial Lipodystrophy
Brief Title: A Study to Examine the Effects of the Leptin Receptor (LEPR) Agonist Antibody REGN4461 in Adult Patients With Familial Partial Lipodystrophy (FPLD)
Acronym: LEAP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R4461-PLD-20100; 2021-000138-33 (EudraCT Number)
Record Dates: First submitted 2021-10-12; First posted 2021-10-22 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-08

CONDITIONS: Familial Partial Lipodystrophy; Metabolic Abnormalities
MeSH Terms: conditions — Lipodystrophy, Familial Partial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Arm 1 (Experimental): Randomized to placebo for 12 weeks and then crossover to REGN4461 for 12 weeks
  Interventions: Drug: REGN4461; Drug: Matching Placebo
- Study Arm 2 (Experimental): Randomized to receive REGN4461 for 24 weeks
  Interventions: Drug: REGN4461

INTERVENTIONS:
Drug: REGN4461 — Intravenous (IV) infusion loading dose followed by subcutaneous (SC) injection weekly (QW).
  Other Names: mibavademab
Drug: Matching Placebo — Intravenous (IV) infusion loading dose followed by subcutaneous (SC) injection weekly (QW).
  Arms: Study Arm 1

SUMMARY:
Two cohorts are being studied based on leptin levels. Cohort A is composed of patients with baseline leptin <8.0 ng/mL and Cohort B is composed of patients with baseline leptin 8.0 to ≤20.0 ng/mL

The primary objectives will be evaluated for patients in Cohort A only:

* To evaluate the effect of REGN4461 on fasting triglycerides (TG) in patients with elevated baseline fasting TG
* To evaluate the effect of REGN4461 on hyperglycemia in patients with elevated baseline Hemoglobin A1c (HbA1c)

The following secondary objectives of the study will be evaluated for Cohort B and for the combined set of Cohorts A plus B:

* To evaluate the effect of REGN4461 on fasting TG levels in patients with hypertriglyceridemia
* To evaluate the effect of REGN4461 on glycemic control in patients with hyperglycemia

The following secondary objectives of the study will be evaluated for Cohorts A and B separately, and for the combined set of Cohorts A plus B:

* To evaluate the effect of REGN4461 on liver fat in patients with hepatic steatosis
* To evaluate the effect of REGN4461 on hunger
* To evaluate safety and tolerability of REGN4461
* To characterize the concentration profile of REGN4461 over time
* To assess immunogenicity to REGN4461

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of familial partial lipodystrophy as defined in the protocol
* Fasting leptin level ≤20.0 ng/ml, as determined during the screening period
* Presence of significant metabolic abnormalities related to glucose and triglycerides (TGs) as defined in the protocol
* Stable body weight within the 3 months prior to screening (no gain or loss of >5% current weight)
* Stable diet during the past 3 months defined as no major change in macronutrient composition (eg, starting or stopping diets such as Atkins, Paleo, Vegetarianism, Veganism)
* No clinically meaningful change in medication regimen in the 3 months prior to screening as defined in the protocol

Key Exclusion Criteria:

* Treatment with metreleptin within 3 months of the screening visit
* Patients with a diagnosis of generalized lipodystrophy
* Patients with a diagnosis of acquired lipodystrophy
* Pregnant or breastfeeding women

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (8):
- United States (5):
  - Excel Medical Clinical Trials - A Flourish Research Site, Boca Raton, Florida
  - National Institute of Health, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
- ICAN, Institute of Cardiometabolism and Nutrition, Paris, France
- Complexo Hospitalario Universitario de Santiago-Hospital Médico-Cirúrxico de Conxo, Santiago de Compostela, Galicia, Spain
- Ege University Faculty of Medicine, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., Food and Drug Administration (FDA), European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

REFERENCES:
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 66 participants were screened, of whom 20 were randomized and received study treatment.
Groups:
- Arm 1 Cohort A: Placebo to REGN4461; Arm 1 Cohort B: Placebo to REGN4461: Participants randomized to Arm 1 received placebo for 12 weeks during the DBTP followed by crossover to REGN4461 treatment for 12 weeks during the SBTP.
- Arm 2 Cohort A: REGN4461 to REGN4461; Arm 2 Cohort B: REGN4461 to REGN4461: Participants randomized to Arm 2 received REGN4461 treatment for 12 weeks during the DBTP followed by an additional 12 weeks of REGN4461 treatment during the SBTP.
Period: Overall Study
Arm/Group | Arm 1 Cohort A: Placebo to REGN4461 | Arm 2 Cohort A: REGN4461 to REGN4461 | Arm 1 Cohort B: Placebo to REGN4461 | Arm 2 Cohort B: REGN4461 to REGN4461
Started (Randomized) | 6 | 6 | 4 | 4
Completed Treatment During DBTP (Double-blind Treatment Period (DBTP)) | 5 (1 participant prematurely discontinued before completing the DBTP at the request of the sponsor due to the early study termination.) | 6 | 4 | 4
Completed Treatment During SBTP (Single-blind Treatment Period (SBTP)) | 5 | 5 (1 participant prematurely discontinued study treatment before completing SBTP at the request of the sponsor due to the early study termination.) | 3 (1 participant completed the DBTP but was prematurely discontinued before entering the SBTP at the request of the sponsor due to the early study termination.) | 4
Completed (Completed study All 20 participants were considered to have completed the study, including the 3 participants who were discontinued at the request of the sponsor during treatment) | 6 | 6 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The double-blind safety analysis set (DB SAF) included all randomized participants who received any study drug during the double-blind treatment period (DBTP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Cohort A: Placebo to REGN4461 | Arm 2 Cohort A: REGN4461 to REGN4461 | Arm 1 Cohort B: Placebo to REGN4461 | Arm 2 Cohort B: REGN4461 to REGN4461 | Total
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (16.79) | 43.8 (13.47) | 48.0 (11.97) | 40.3 (12.82) | 43.0 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 3 | 4 | 18
  Male | 1 | 0 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 4 | 4 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 3 | 3 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Fasting Triglycerides Serum Concentration [Geometric Mean (Full Range); unit: milligrams per deciliter (mg/dL)] | 1100.9 [405 to 5681] | 737.8 [308 to 2487] | 675.0 [426 to 1534] | 336.2 [150 to 1376] | 698.3 [150 to 5681]
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 8.8 (1.62) | 8.2 (1.76) | 6.9 (0.91) | 8.6 (2.06) | 8.2 (1.68)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 in Fasting Serum Triglyceride (TG) (Cohort A)
Description: Percentage change in fasting serum TG was reported for participants with elevated baseline fasting TG (> 200 mg/dL) and with baseline leptin < 8.0 ng/mL (Cohort A).
Time Frame: Baseline to week 12
Population: The Full Analysis Set (FAS) included all randomized participants who received any study drug in the double-blind treatment period (DBTP) and had at least 1 post-baseline assessment. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm 1 Cohort A: Placebo to REGN4461 | Arm 2 Cohort A: REGN4461 to REGN4461
Number analyzed (Participants) | 5 | 6
percent change | -11.30 (46.306) | -38.97 (16.998)

2. Primary Outcome: Change From Baseline to Week 12 in Hemoglobin A1c (HbA1c) (Cohort A)
Description: Change in HbA1c was reported for participants with elevated baseline HbA1c (> 7.0%) and with baseline leptin < 8.0 ng/mL (Cohort A).
Time Frame: Baseline to week 12
Population: The FAS included all randomized participants who received any study drug in the DBTP and had at least 1 post-baseline assessment. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Arm 1 Cohort A: Placebo to REGN4461 | Arm 2 Cohort A: REGN4461 to REGN4461
Number analyzed (Participants) | 4 | 5
percentage of glycated hemoglobin | -0.05 (0.451) | -1.08 (1.108)

3. Secondary Outcome: Percent Change From Baseline to Week 12 in Fasting Serum TG (Cohorts B and A + B)
Description: Percent change in fasting serum TG was reported for participants with elevated baseline fasting TG (>200 mg/dL) in Cohort B and Cohorts A + B.
Time Frame: Baseline to week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Arm 1 Combined Cohort A + B: Placebo to REGN4461: "Arm 1 Cohort A" and "Arm 1 Cohort B" combined
- Arm 2 Combined Cohort A + B: REGN4461 to REGN4461: "Arm 2 Cohort A" and "Arm 2 Cohort B" combined
Arm/Group | Arm 1 Cohort B: Placebo to REGN4461 | Arm 2 Cohort B: REGN4461 to REGN4461 | Arm 1 Combined Cohort A + B: Placebo to REGN4461 | Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 4 | 4 | 9 | 10
percent change | 36.78 (44.863) | -35.59 (8.754) | 10.07 (49.689) | -37.62 (13.752)

4. Secondary Outcome: Change From Baseline to Week 12 in HbA1c (Cohorts B and A + B)
Description: Change in HbA1c was reported for participants with elevated baseline HbA1c (>7.0%) in Cohort B and Cohorts A + B.
Time Frame: Baseline to week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Arm 1 Cohort B: Placebo to REGN4461 | Arm 2 Cohort B: REGN4461 to REGN4461 | Arm 1 Combined Cohort A + B: Placebo to REGN4461 | Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 2 | 3 | 6 | 8
percentage of glycated hemoglobin | -0.20 (0.283) | -0.90 (0.964) | -0.10 (0.379) | -1.01 (0.988)

5. Secondary Outcome: Percent Change From Baseline to Weeks 12 and 24 in Fasting Serum TG (Study Arm 1)
Description: Percent change in fasting serum TG was reported for participants in Study Arm 1.
Time Frame: Baseline, Week 12, Week 24
Population: The FAS included all randomized participants who received any study drug in the DBTP and had at least 1 post-baseline assessment. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure, and "Number analyzed" is the number of participants evaluated at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm 1 Cohort A: Placebo to REGN4461 | Arm 1 Cohort B: Placebo to REGN4461 | Arm 1 Combined Cohort A + B: Placebo to REGN4461
Number analyzed (Participants) | 5 | 4 | 9
percent change
  Week 12 | -11.30 (46.306) | 36.78 (44.863) | 10.07 (49.689)
  Week 24: number analyzed (Participants) | 5 | 2 | 7
  Week 24 | -29.79 (35.109) | -8.96 (13.673) | -23.84 (30.923)

6. Secondary Outcome: Percent Change From Baseline to Weeks 12 and 24 in Fasting Serum TG (Study Arm 2)
Description: Percent change in fasting serum TG was reported for participants in Study Arm 2.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm 2 Cohort A: REGN4461 to REGN4461 | Arm 2 Cohort B: REGN4461 to REGN4461 | Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 6 | 4 | 10
percent change
  Week 12 | -38.97 (16.998) | -35.59 (8.754) | -37.62 (13.752)
  Week 24: number analyzed (Participants) | 4 | 4 | 8
  Week 24 | -30.77 (48.883) | -5.30 (51.158) | -18.04 (48.282)

7. Secondary Outcome: Change From Baseline to Weeks 12 and 24 in HbA1c (Study Arm 1)
Description: Change from baseline in HbA1c was reported for participants in Study Arm 1.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Arm 1 Cohort A: Placebo to REGN4461 | Arm 1 Cohort B: Placebo to REGN4461 | Arm 1 Combined Cohort A + B: Placebo to REGN4461
Number analyzed (Participants) | 5 | 4 | 9
percentage of glycated hemoglobin
  Week 12 | -0.10 (0.406) | 0.13 (0.427) | 0.00 (0.406)
  Week 24: number analyzed (Participants) | 5 | 3 | 8
  Week 24 | -0.78 (0.694) | 0.13 (0.802) | -0.44 (0.826)

8. Secondary Outcome: Change From Baseline to Weeks 12 and 24 in HbA1c (Study Arm 2)
Description: Change from baseline in HbA1c was reported for participants in Study Arm 2.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Arm 2 Cohort A: REGN4461 to REGN4461 | Arm 2 Cohort B: REGN4461 to REGN4461 | Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 6 | 4 | 10
percentage of glycated hemoglobin
  Week 12 | -0.92 (1.068) | -0.78 (0.826) | -0.86 (0.931)
  Week 24: number analyzed (Participants) | 5 | 4 | 9
  Week 24 | -0.98 (1.357) | -0.50 (1.068) | -0.77 (1.188)

9. Secondary Outcome: Change From Baseline to Weeks 12 and 24 in Fasting Glucose (Study Arm 1)
Description: Change from baseline in fasting glucose was reported for participants in Study Arm 1.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Arm 1 Cohort A: Placebo to REGN4461 | Arm 1 Cohort B: Placebo to REGN4461 | Arm 1 Combined Cohort A + B: Placebo to REGN4461
Number analyzed (Participants) | 5 | 4 | 9
milligrams per deciliter (mg/dL)
  Week 12 | 4.8 (29.55) | 0.0 (60.37) | 2.7 (42.54)
  Week 24: number analyzed (Participants) | 5 | 2 | 7
  Week 24 | 7.2 (29.65) | -15.5 (6.36) | 0.7 (26.75)

10. Secondary Outcome: Change From Baseline to Weeks 12 and 24 in Fasting Glucose (Study Arm 2)
Description: Change from baseline in fasting glucose was reported for participants in Study Arm 2.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 2 Cohort A: REGN4461 to REGN4461 | Arm 2 Cohort B: REGN4461 to REGN4461 | Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 6 | 4 | 10
mg/dL
  Week 12 | -5.2 (36.55) | -19.5 (22.87) | -10.9 (31.17)
  Week 24: number analyzed (Participants) | 4 | 4 | 8
  Week 24 | 1.8 (26.35) | -12.3 (58.59) | -5.3 (42.71)

11. Secondary Outcome: Percent Change From Baseline to Weeks 12 and 24 in Liver Fat Magnetic Resonance Imaging-derived Proton Density Fat Fraction (MRI-PDFF) (Study Arm 1)
Description: Percent change from baseline in MRI-PDFF was reported for participants with baseline MRI-PDFF ≥8.5% in Study Arm 1.
Time Frame: Baseline, Week 12, Week 24
Population: The FAS included all randomized participants who received any study drug in the DBTP and had at least 1 post-baseline assessment. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure with baseline MRI-PDFF ≥8.5%, and "Number analyzed" is the number of participants evaluated at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm 1 Cohort A: Placebo to REGN4461 | Arm 1 Cohort B: Placebo to REGN4461 | Arm 1 Combined Cohort A + B: Placebo to REGN4461
Number analyzed (Participants) | 3 | 2 | 5
percent change
  Week 12 | -11.44 (18.576) | -0.74 (9.919) | -7.16 (15.214)
  Week 24: number analyzed (Participants) | 2 | 1 | 3
  Week 24 | -47.21 (22.176) | 44.81 (NA) — SD not calculable with n=1 | -16.54 (55.394)

12. Secondary Outcome: Percent Change From Baseline to Weeks 12 and 24 in Liver Fat MRI-PDFF (Study Arm 2)
Description: Percent change from baseline in MRI-PDFF was reported for participants with baseline liver fat MRI-PDFF ≥8.5% in Study Arm 2.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arm 2 Cohort A: REGN4461 to REGN4461 | Arm 2 Cohort B: REGN4461 to REGN4461 | Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 4 | 4 | 8
percent change
  Week 12 | -17.05 (25.788) | -18.80 (17.300) | -17.92 (20.351)
  Week 24: number analyzed (Participants) | 4 | 3 | 7
  Week 24 | -24.33 (27.151) | -19.53 (19.324) | -22.27 (22.353)

13. Secondary Outcome: Change From Baseline to Weeks 12 and 24 on the Daily Lipodystrophy Hunger Questionnaire - Highest Hunger Score
Description: The daily lipodystrophy hunger questionnaire was developed to assess hunger related behaviors among patients with lipodystrophy. The highest hunger score asked participants to rate their highest hunger that day on a scale from 0 to 4, with higher scores representing the higher perceived hunger. A negative change from baseline indicated a reduction in perceived hunger.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 Cohort A: Placebo to REGN4461 | Arm 2 Cohort A: REGN4461 to REGN4461 | Arm 1 Cohort B: Placebo to REGN4461 | Arm 2 Cohort B: REGN4461 to REGN4461 | Arm 1 Combined Cohort A + B: Placebo to REGN4461 | Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 10 | 10
score on a scale
  Week 12 | -0.060 (0.9009) | -0.538 (0.4679) | -0.240 (0.2483) | -0.415 (0.7539) | -0.132 (0.6929) | -0.489 (0.5614)
  Week 24: number analyzed (Participants) | 5 | 5 | 3 | 4 | 8 | 9
  Week 24 | -0.330 (0.3684) | -0.018 (0.6228) | -0.383 (0.1550) | -0.285 (0.6180) | -0.350 (0.2919) | -0.137 (0.5975)

14. Secondary Outcome: Change From Baseline to Weeks 12 and 24 on the Daily Lipodystrophy Hunger Questionnaire - Lowest Hunger Score
Description: The daily lipodystrophy hunger questionnaire was developed to assess hunger related behaviors among patients with lipodystrophy. The lowest hunger score asked participants to rate their lowest hunger that day on a scale from 0 to 4, with higher scores indicating higher perceived hunger. A negative change from baseline score indicated a reduction in perceived lowest hunger.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 Cohort A: Placebo to REGN4461 | Arm 2 Cohort A: REGN4461 to REGN4461 | Arm 1 Cohort B: Placebo to REGN4461 | Arm 2 Cohort B: REGN4461 to REGN4461 | Arm 1 Combined Cohort A + B: Placebo to REGN4461 | Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 10 | 10
score on a scale
  Week 12 | 0.185 (0.8013) | -0.475 (0.4630) | -0.338 (0.4287) | -0.173 (0.3625) | -0.024 (0.7006) | -0.354 (0.4328)
  Week 24: number analyzed (Participants) | 5 | 5 | 3 | 4 | 8 | 9
  Week 24 | -0.128 (0.0622) | 0.046 (0.6776) | -0.103 (0.2230) | 0.308 (0.9603) | -0.119 (0.1288) | 0.162 (0.7710)

15. Secondary Outcome: Change From Baseline to Weeks 12 and 24 on the Daily Lipodystrophy Hunger Questionnaire - Felt Hungry Score
Description: The daily lipodystrophy hunger questionnaire was developed to assess hunger related behaviors among participants with lipodystrophy. The felt hungry score asked how much time participants felt hunger that day on a scale from 0 to 4, with higher scores indicating more time feeling hungry. A negative change from baseline score indicated a reduction in time spent feeling hungry.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 Cohort A: Placebo to REGN4461 | Arm 2 Cohort A: REGN4461 to REGN4461 | Arm 1 Cohort B: Placebo to REGN4461 | Arm 2 Cohort B: REGN4461 to REGN4461 | Arm 1 Combined Cohort A + B: Placebo to REGN4461 | Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 10 | 10
score on a scale
  Week 12 | 0.248 (0.8642) | -0.550 (0.5334) | -0.168 (0.2900) | 0.008 (0.9139) | 0.082 (0.6993) | -0.327 (0.7206)
  Week 24: number analyzed (Participants) | 5 | 5 | 3 | 4 | 8 | 9
  Week 24 | 0.016 (0.3932) | 0.120 (0.4374) | -0.183 (0.0603) | -0.138 (0.6595) | -0.059 (0.3163) | 0.006 (0.5265)

16. Secondary Outcome: Change From Baseline to Weeks 12 and 24 on the Daily Lipodystrophy Hunger Questionnaire - Fullness Score
Description: The daily lipodystrophy hunger questionnaire was developed to assess hunger related behaviors among patients with lipodystrophy. The fullness score asked participants to rate how often they felt full after eating that day on a scale from 0 to 4, with higher scores indicating higher feeling of fullness. A negative change from baseline indicated a reduced feeling of fullness.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 Cohort A: Placebo to REGN4461 | Arm 2 Cohort A: REGN4461 to REGN4461 | Arm 1 Cohort B: Placebo to REGN4461 | Arm 2 Cohort B: REGN4461 to REGN4461 | Arm 1 Combined Cohort A + B: Placebo to REGN4461 | Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 10 | 10
score on a scale
  Week 12 | 0.063 (1.1988) | -0.267 (0.5381) | -1.180 (0.3764) | -0.535 (0.5736) | -0.434 (1.1216) | -0.374 (0.5383)
  Week 24: number analyzed (Participants) | 5 | 5 | 3 | 4 | 8 | 9
  Week 24 | -0.182 (0.6474) | 0.012 (0.6474) | -1.193 (0.6630) | -0.178 (0.8032) | -0.561 (0.7994) | -0.072 (0.6793)

17. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: Up to Day 169
Population: The DB SAF included all participants who received any double-blind study drug in DBTP. The single-blind safety analysis set (SB SAF) included all randomized participants who received any single-blind study drug in the single-blind treatment period (SBTP).
Measure: Count of Participants; unit: Participants
Groups:
- DBTP Arm 1 Cohort A: Placebo; DBTP Arm 1 Cohort B: Placebo: Participants randomized to Arm 1 received placebo for 12 weeks during the DBTP.
- DBTP Arm 2 Cohort A: REGN4461; DBTP Arm 2 Cohort B: REGN4461: Participants randomized to Arm 2 received REGN4461 treatment for 12 weeks during the DBTP.
- DBTP Arm 1 Combined Cohort A + B: Placebo: DBTP "Arm 1 Cohort A" and "Arm 1 Cohort B" combined
- DBTP Arm 2 Combined Cohort A + B: REGN4461: DBTP "Arm 2 Cohort A" and "Arm 2 Cohort B" combined
- SBTP Arm 1 Cohort A: Placebo to REGN4461; SBTP Arm 1 Cohort B: Placebo to REGN4461: Participants randomized to Arm 1 received placebo for 12 weeks during the DBTP followed by crossover to REGN4461 treatment for 12 weeks during the SBTP.
- SBTP Arm 2 Cohort A: REGN4461 to REGN4461; SBTP Arm 2 Cohort B: REGN4461 to REGN4461: Participants randomized to Arm 2 received REGN4461 treatment for 12 weeks during the DBTP followed by an additional 12 weeks of REGN4461 treatment during the SBTP.
- SBTP Arm 1 Combined Cohort A + B: Placebo to REGN4461: SBTP "Arm 1 Cohort A" and "Arm 1 Cohort B" combined
- SBTP Arm 2 Combined Cohort A + B: REGN4461 to REGN4461: SBTP "Arm 2 Cohort A" and "Arm 2 Cohort B" combined
Arm/Group | DBTP Arm 1 Cohort A: Placebo | DBTP Arm 2 Cohort A: REGN4461 | DBTP Arm 1 Cohort B: Placebo | DBTP Arm 2 Cohort B: REGN4461 | DBTP Arm 1 Combined Cohort A + B: Placebo | DBTP Arm 2 Combined Cohort A + B: REGN4461 | SBTP Arm 1 Cohort A: Placebo to REGN4461 | SBTP Arm 2 Cohort A: REGN4461 to REGN4461 | SBTP Arm 1 Cohort B: Placebo to REGN4461 | SBTP Arm 2 Cohort B: REGN4461 to REGN4461 | SBTP Arm 1 Combined Cohort A + B: Placebo to REGN4461 | SBTP Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 10 | 10 | 5 | 6 | 3 | 4 | 8 | 10
Participants | 4 | 5 | 4 | 4 | 8 | 9 | 3 | 5 | 3 | 4 | 6 | 9

18. Secondary Outcome: Concentrations of REGN4461 in Serum
Time Frame: Weeks 0, 1, 2, 3, 4, 5, 6, 9, 12, 13, 14, 15, 16, 17, 18, 21, 28, 32 and 36. Weeks 0 and 12 collected pre- and post-dose. All other time points were only pre-dose.
Population: The PK analysis set was defined as all randomized participants who received any study drug and have at least 1 non-missing measurement of REGN4461 concentration following the first dose of study drug. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure, and "Number analyzed" is the number of participants evaluated at each time point.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Arm 1 Combined Cohort A + B: Placebo to REGN4461 | Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 10 | 10
milligrams per liter (mg/L)
  Week 0 (pre-dose) | 0 (0) | 0 (0)
  Week 0 (post-dose) | 0 (0) | 232 (83.8)
  Week 1 (pre-dose): number analyzed (Participants) | 9 | 8
  Week 1 (pre-dose) | 0 (0) | 64.3 (24.9)
  Week 2 (pre-dose): number analyzed (Participants) | 9 | 10
  Week 2 (pre-dose) | 0 (0) | 52.5 (13.3)
  Week 3 (pre-dose): number analyzed (Participants) | 10 | 8
  Week 3 (pre-dose) | 0 (0) | 60.2 (19.0)
  Week 4 (pre-dose): number analyzed (Participants) | 8 | 10
  Week 4 (pre-dose) | 0 (0) | 58.8 (23.8)
  Week 5 (pre-dose) | 0 (0) | 62.0 (36.1)
  Week 6 (pre-dose) | 0 (0) | 68.8 (38.8)
  Week 9 (pre-dose): number analyzed (Participants) | 10 | 9
  Week 9 (pre-dose) | 0 (0) | 79.6 (49.2)
  Week 12 (pre-dose): number analyzed (Participants) | 8 | 10
  Week 12 (pre-dose) | 0 (0) | 87.1 (57.8)
  Week 12 (post-dose): number analyzed (Participants) | 8 | 10
  Week 12 (post-dose) | 252 (50.7) | 87.6 (49.7)
  Week 13 (pre-dose): number analyzed (Participants) | 8 | 10
  Week 13 (pre-dose) | 62.4 (17.5) | 97.6 (68.6)
  Week 14 (pre-dose): number analyzed (Participants) | 8 | 10
  Week 14 (pre-dose) | 56.6 (17.6) | 92.8 (68.0)
  Week 15 (pre-dose): number analyzed (Participants) | 8 | 10
  Week 15 (pre-dose) | 64.2 (29.6) | 90.5 (59.1)
  Week 16 (pre-dose): number analyzed (Participants) | 8 | 10
  Week 16 (pre-dose) | 68.8 (24.3) | 103 (76.4)
  Week 17 (pre-dose): number analyzed (Participants) | 8 | 10
  Week 17 (pre-dose) | 73.4 (30.8) | 92.1 (73.3)
  Week 18 (pre-dose): number analyzed (Participants) | 8 | 10
  Week 18 (pre-dose) | 75.1 (27.1) | 95.0 (79.3)
  Week 21 (pre-dose): number analyzed (Participants) | 8 | 9
  Week 21 (pre-dose) | 89.3 (40.0) | 72.9 (51.4)
  Week 28 (pre-dose) | 10.9 (12.0) | 16.0 (23.4)
  Week 32 (pre-dose): number analyzed (Participants) | 9 | 10
  Week 32 (pre-dose) | 0.0663 (0.0705) | 0.189 (0.281)
  Week 36 (pre-dose): number analyzed (Participants) | 9 | 10
  Week 36 (pre-dose) | 0.0110 (0.0330) | 0.0373 (0.0788)

19. Secondary Outcome: Number of Participants With Treatment-emergent Anti-drug Antibody (ADA) Response
Time Frame: Up to Day 281
Population: The ADA analysis set included all treated participants who received any amount of study drug and had at least one non-missing anti-drug antibody result following the first dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Combined Cohort A + B: Placebo to REGN4461 | Arm 2 Combined Cohort A + B: REGN4461 to REGN4461
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to day 281 (end of study)
Arm/Group | DBTP Arm 1 Cohort A: Placebo | DBTP Arm 2 Cohort A: REGN4461 | DBTP Arm 1 Cohort B: Placebo | DBTP Arm 2 Cohort B: REGN4461 | SBTP Arm 1 Cohort A: Placebo to REGN4461 | SBTP Arm 2 Cohort A: REGN4461 to REGN4461 | SBTP Arm 1 Cohort B: Placebo to REGN4461 | SBTP Arm 2 Cohort B: REGN4461 to REGN4461
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/4 | 0/5 | 0/6 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 1/4 | 0/4 | 1/5 | 1/6 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 4/4 | 4/4 | 3/5 | 5/6 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBTP Arm 1 Cohort A: Placebo (N=6) | DBTP Arm 2 Cohort A: REGN4461 (N=6) | DBTP Arm 1 Cohort B: Placebo (N=4) | DBTP Arm 2 Cohort B: REGN4461 (N=4) | SBTP Arm 1 Cohort A: Placebo to REGN4461 (N=5) | SBTP Arm 2 Cohort A: REGN4461 to REGN4461 (N=6) | SBTP Arm 1 Cohort B: Placebo to REGN4461 (N=3) | SBTP Arm 2 Cohort B: REGN4461 to REGN4461 (N=4)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBTP Arm 1 Cohort A: Placebo (N=6) | DBTP Arm 2 Cohort A: REGN4461 (N=6) | DBTP Arm 1 Cohort B: Placebo (N=4) | DBTP Arm 2 Cohort B: REGN4461 (N=4) | SBTP Arm 1 Cohort A: Placebo to REGN4461 (N=5) | SBTP Arm 2 Cohort A: REGN4461 to REGN4461 (N=6) | SBTP Arm 1 Cohort B: Placebo to REGN4461 (N=3) | SBTP Arm 2 Cohort B: REGN4461 to REGN4461 (N=4)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plicated tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain fog (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mononeuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Poor quality sleep (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (10) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbohydrate antigen 19-9 increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the Sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT05088460/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT05088460/SAP_001.pdf